CLINICAL TRIAL: NCT02520934
Title: Evaluation of Combination Therapy With Miglustat and Enzyme Replacement Therapy on Gaucher Disease Type IIIB
Brief Title: Miglustat on Gaucher Disease Type IIIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503076MIPD
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Gaucher Disease
Keywords: Enzyme Replacement Therapy; Miglustat; Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case_Miglustat (Experimental): Besides regular ERT, patients in this group also need to take Miglustat for 24 months.
  Interventions: Drug: Miglustat; Drug: ERT
- Control (No Intervention): Patients will be tested for their pupil cycle time.

INTERVENTIONS:
Drug: Miglustat — combine miglustat and ERT to see if neurologic manifestations can be improved
  Other Names: Zavesca
  Arms: Case_Miglustat
Drug: ERT — enzyme replacement therapy
  Arms: Case_Miglustat

SUMMARY:
evaluate the combination therapy with Miglustat and enzyme replacement therapy (ERT) on Gaucher disease

DETAILED DESCRIPTION:
understand if Miglustat (glucosylceramide synthase inhibitor) could improve neuropathy in patients with Gaucher disease

ELIGIBILITY:
Case_Miglustat

Inclusion Criteria:

1. Confirmed diagnosis of Gaucher Disease: blood test shown lack of beta- glucocerebrosidase, and found L444P homozygous on GBA gene.
2. Aged 6 years old or above.
3. Already have regular ERT (30-120 IU/kg/ every 2 weeks) at least a year; dosage and frequency of ERT had not been changed in recent 3 months.

Exclusion Criteria:

1. History of tremor and abnormal extremities perception ( pain, numbness, tingle etc.)
2. Abnormal kidney function.
3. Pregnant or plan to have a baby ( potentially pregnant patient need to be transferred to gynecologist for the test and promise to have proper contraception measures).
4. Allergic to Miglustat.

Control_normal Inclusion Criteria

1. Age 6-18 years
2. No significant physical, mental, or psychiatric problems

Exclusion criteria

1. Children with eye disease (not include myopia, hyperopia, Astigmatism)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Improve in Purdue Pegboard test speed | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan